CLINICAL TRIAL: NCT03062865
Title: "ART REGISTRY : Rheumatoid Arthritis and Anti-TNF"
Brief Title: French National Registry: ART REGISTRY (Observational Study)
Acronym: ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Societe Francaise de Rhumatologie (Other)
Responsible Party: Sponsor
Other Study IDs: ART
Record Dates: First submitted 2017-01-13; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: RheumatoId Arthritis
Keywords: Rheumatoid arthritis (RA); TNF-alpha inhibitors
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
Rheumatoid arthritis (RA) is a complex and multifactorial autoimmune disease. The biological treatments that are currently available for the treatment of RA are the TNF-alpha inhibitors. Tumor necrosis factor (TNF) is a dominant cytokine in the inflammatory process of rheumatoid arthritis. The anti-TNFs were the first to enter the market, and they revolutionised the prognoses of patients with RA. They remain the most common first-line biotherapy and are the most used at this time.

The French Society of Rheumatologists intends to coordinate a prospective national registry study for this follow-up.

This registry will include 1500 RA patients from the start of treatment with anti-TNF-α and then followed for 5 years, regardless of the therapeutic modifications occurring thereafter.

This registry is an observational, multicentre, longitudinal, prospective registry study The objectives of this registry is to contribute 1) to evaluate the therapeutic management of patients; and 2) to improve this therapeutic management.

DETAILED DESCRIPTION:
Design: Observational, multicentre, longitudinal, prospective registry Primary objective: To evaluate the real life efficacy and safety of anti-TNF inhibitors in patients with RA using a prospective national registry.

Target population: Patients initiating anti-TNF therapy for RA (including infliximab, adalimumab, etanercept, certolizumab and golimumab, and their respective biosimilar according to their arrival on the market) Number of patients and centres : More than 80 centers in France (hospital-based, public and private practice) Recruitment period: 3 years Follow-up: 5 years

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with RA,
* Patient in whom the specialist physician decides to start treatment with an anti-TNF drug, regardless of the treatment line and regardless of the anti-TNF, including infliximab, adalimumab, etanercept, certolizumab and golimumab, and their respective biosimilar according to their arrival on the market
* Clinicians (hospital-based and private practice) who agree to adhere to the yearly renewal of the hospital prescription

Exclusion Criteria:

* Patient already treated by the same anti-TNF in the past (same drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population :
  Patients with rheumatoid arthritis initiating anti-TNF therapy, whatever the treatment line
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-11; Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Drug (anti TNF inhibitors) retention rate | From the beginning of the study until the end of the 5 years follow-up
  Primary outcome will be 5-year drug retention, this rate will be compared between the different drugs to assess real life efficacy of anti-TNF inhibitors in patients with RA

SECONDARY OUTCOMES:
Treatment retention rate on anti-TNF therapy | From the beginning of the study until the end of the 5 years follow-up
  * outcome : 1, 2, 3, 4 and 5-year drug retention rate
  * comparisons : between all the TNF inhibitors
Number of patients receiving each of the drugs | From the beginning of the study until the end of the 5 years follow-up
  Place of anti-TNF agents among the therapeutic choices
- Number and nature of biologics previously received | From the beginning of the study until the end of the 5 years follow-up
  Place of anti-TNF agents among the therapeutic choices
rate of serious and opportunistic infections (overall and subtypes) | From the beginning of the study until the end of the 5 years follow-up
  Safety Outcome
Rate of malignancies (overall and subtypes) | From the beginning of the study until the end of the 5 years follow-up
  Safety Outcome
Rate of cardiovascular events (overall and subtypes) | From the beginning of the study until the end of the 5 years follow-up
  Safety Outcome
rate of serious adverse events (overall and subtypes) | From the beginning of the study until the end of the 5 years follow-up
  Safety Outcome
Rate of surgery and surgical complications (overall and subtypes) | From the beginning of the study until the end of the 5 years follow-up
  Safety Outcome
Comparison with the other french biotherapy registries with similar methodology | From the beginning of the study until the end of the 5 years follow-up
  - comparisons of the following outcomes: drug retention rate, rate of serious infections, rate of malignancies, rate of serious adverse events, rate of cardiovascular events
Establishment of a database accessible to all participating clinicians in the collection for the purpose of making complementary analyses. | From the beginning of the study until the end of the 5 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Raphaele SEROR, Principal Investigator — SFR/AP-HP
Locations (1):
- Hopital Bicêtre, Le Kremlin-Bicêtre, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen Y, Baron G, Hamamouche N, Belkhir R, Miconnet S, Soubrier M, Hostachy C, Thevenot P, Basch A, Truchetet ME, Claudepierre P, Dernis E, Marotte H, Flipo RM, Brocq O, Morel J, Fautrel B, Salliot C, Saraux A, Leske C, Schaeverbeke T, Ravaud P, Mariette X, Ruyssen-Witrand A, Seror R; ART Study Group section sign. Do SMS/e-mail reminders increase influenza vaccination of rheumatoid arthritis patients under anti-TNF: a nested randomized controlled trial in the ART e-cohort. Rheumatology (Oxford). 2025 May 1;64(5):2496-2504. doi: 10.1093/rheumatology/keae599. PMID 39576675